CLINICAL TRIAL: NCT03201874
Title: iCanCope With Sickle Cell Disease: A Mobile Pain Management Intervention for Adolescents
Brief Title: iCanCope With Sickle Cell Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: The Hospital for Sick Children (Other); Emory University (Other); Connecticut Children's Medical Center (Other); University of Mississippi Medical Center (Other); University of Florida (Other); Boston Medical Center (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Tonya Palermo, Professor, Anesthesiology and Pain Medicine, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01HD086978 (NIH)
Record Dates: First submitted 2017-06-23; First posted 2017-06-28 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Control (Active Comparator): In addition to standard medical care, youth in the education control group will be provided with access to a self-guided education study website, which will contain static education about SCD (no self-management skills, goal-setting, or social support content) to access over 8-weeks.
  Interventions: Behavioral: Education
- Pain Self-Management Intervention (Experimental): In addition to standard medical SCD care, youth in the pain self-management intervention group will receive the iCanCope with SCD mobile intervention including goal-setting, peer social support, and pain self-management skills over a period of 8 weeks.
  Interventions: Behavioral: Pain self-management; Behavioral: Education

INTERVENTIONS:
Behavioral: Pain self-management — The program is designed to enhance self-efficacy. The app will guide youth in setting structured and personalized goals aimed at improving their pain and functioning. The pain self-management skills will include personalized CBT-based coping skills including deep breathing, relaxation, and cognitive skills (e.g., staying positive). The app will provide in-the-moment access to pain coping strategies to promote positive changes in mood, behavior, and pain.
  Arms: Pain Self-Management Intervention
Behavioral: Education — Education about sickle cell disease to increase disease knowledge

SUMMARY:
The project will test a tailored web and smartphone-based application (iCanCope with SCD) to improve pain self-management and functioning in youth (aged 12-18) with sickle cell disease. The program will include goal setting, peer-based social support, and pain self-management training. The investigators will determine initial program effectiveness through a pilot three-site randomized controlled trial in 160 youth randomized to treatment compared to attention control.

DETAILED DESCRIPTION:
Cognitive-behavioral therapies (CBT) that promote pain self-management can lead to symptom reduction, improved quality of life, and decreased healthcare use. However, most people with SCD do not receive CBT-based treatment due to barriers such as poor accessibility, limited availability of professionals, and high costs. First, the investigators plan to apply a user-centered design approach to develop and refine the iCanCope with SCD program. Second, program feasibility and initial program effectiveness will be determined through a pilot three-site randomized controlled trial. The investigators will determine study accrual and dropout rates as well as levels of patient acceptability and engagement. Preliminary effectiveness will be determined in youth receiving treatment compared to attention control on a range of physical, behavioral, and psychosocial outcomes assessed at post-treatment and 6-month follow-up. Third, moderators and mediators of treatment effect will be tested by examining whether differences in self-efficacy and patient activation predict changes in pain and functioning. These results will enable a future full-scale randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* aged between 12-18 years
* diagnosed with any type of SCD
* able to speak and read English
* score at least 4 (indicating some days with pain interference over the past month) on the Sickle Cell Pain Burden Interview
* willing and able to complete online measures

Exclusion Criteria:

* significant cognitive limitations that would impair their ability to use and understand the iCanCope with SCD program, as per their healthcare provider or parent
* have previously received more than 4 sessions of outpatient psychological therapy for pain management in the 6 months prior to the time of screening.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonya M Palermo, PhD, Principal Investigator — Seattle Children's Hospital
Locations (4):
- United States (3):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Emory University, Atlanta, Georgia
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palermo TM, Srinakarin K, Zhou C, Lalloo C, Dampier C, Zempsky WT, Badawy SM, Bakshi N, Ko YJ, Nishat F, Stinson JN. Moderators of digital cognitive-behavioral therapy for youth with sickle cell disease pain: secondary analysis of a randomized controlled trial. Pain. 2025 Mar 13;166(9):e233-e243. doi: 10.1097/j.pain.0000000000003583. PMID 40839690
- [Derived] Palermo TM, Lalloo C, Zhou C, Dampier C, Zempsky W, Badawy SM, Bakshi N, Ko YJ, Nishat F, Stinson JN. A cognitive-behavioral digital health intervention for sickle cell disease pain in adolescents: a randomized, controlled, multicenter trial. Pain. 2024 Jan 1;165(1):164-176. doi: 10.1097/j.pain.0000000000003009. Epub 2023 Sep 21. PMID 37733479
- [Derived] Lalloo C, Nishat F, Zempsky W, Bakshi N, Badawy S, Ko YJ, Dampier C, Stinson J, Palermo TM. Characterizing User Engagement With a Digital Intervention for Pain Self-management Among Youth With Sickle Cell Disease and Their Caregivers: Subanalysis of a Randomized Controlled Trial. J Med Internet Res. 2022 Aug 30;24(8):e40096. doi: 10.2196/40096. PMID 36040789

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants refers to dyads (parents and adolescents). Enrollment and randomization assignment was by dyad. Indicated in the comments is the number of parents and adolescents.
  26 participants gave consent for did not complete the pre-treatment assessment. Participants were not randomized and assigned to groups. They did not complete baseline.
Period: Baseline
Arm/Group | Education Control | Pain Self-Management Intervention
Started (Parents started Education Control: 54, Adolescents started Education Control: 54, Parents started Pain Self-Management Intervention: 56, Adolescents started Pain Self-Management Intervention: 57) | 54 | 57
Completed (Parents completed Education Control: 50, Adolescents completed Education Control: 54, Parents completed Pain Self-Management Intervention: 55, Adolescents completed Pain Self-Management Intervention: 57) | 54 | 57
Not Completed | 0 | 0
Period: Post-Treatment (12 Weeks)
Arm/Group | Education Control | Pain Self-Management Intervention
Started (Parents started Education Control: 51, Adolescents started Education Control: 54, Parents started Pain Self-Management Intervention: 56, Adolescents started Pain Self-Management Intervention: 57) | 54 | 57
Completed (Parents completed Education Control: 43, Adolescents completed Education Control: 50, Parents completed Pain Self-Management Intervention: 43, Adolescents completed Pain Self-Management Intervention: 52) | 50 | 52
Not Completed | 4 | 5
Not completed — Declined due to lack of time/interest or could not be reached | 4 | 5
Period: Follow-up (26 Weeks)
Arm/Group | Education Control | Pain Self-Management Intervention
Started (Parents started Education Control: 51, Adolescents started Education Control: 54, Parents started Pain Self-Management Intervention: 56, Adolescents started Pain Self-Management Intervention: 57) | 54 | 57
Completed (Parents completed Education Control: 44, Adolescents completed Education Control: 49, Parents completed Pain Self-Management Intervention: 41, Adolescents completed Pain Self-Management Intervention: 49) | 49 | 49
Not Completed | 5 | 8
Not completed — Declined due to lack of time/interest or could not be reached | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education Control | Pain Self-Management Intervention | Total
Number analyzed (Participants) | 54 | 57 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (1.9) | 14.9 (2.0) | 14.8 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 23 | 23 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 44 | 47 | 91
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 51 | 98
  White | 0 | 0 | 0
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 6 | 2 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 16 | 11 | 27
  United States | 38 | 46 | 84
SCD genotype [Count of Participants; unit: Participants] — Clinician diagnosis of type of SCD
  Participants
    SS | 33 | 36 | 69
    SC | 14 | 12 | 26
    S Beta Thal + | 3 | 3 | 6
    S Beta Thal o | 2 | 3 | 5
    Unknown/Missing | 2 | 3 | 5
Currently taking hydroxyurea [Count of Participants; unit: Participants]
  Yes | 34 | 41 | 75
  No | 18 | 15 | 33
  Missing | 2 | 1 | 3
Receiving regular blood transfusions [Count of Participants; unit: Participants]
  Yes | 5 | 8 | 13
  No | 47 | 47 | 94
  Missing | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pain Diary - Average Daily Pain
Description: App diary using an 11-point numerical rating scale for pain intensity for 7 days Scores range from 0-10 where higher scores indicate a worse outcome
Time Frame: Baseline,12 weeks, and 26 weeks
Population: At Post-Treatment 9 subjects (4 Education Control and 5 Pain Self-Management Intervention) declined to participate or could not be reached. At Follow-up 13 subjects declined to participate or could not be reached (5 Education Control and 8 Pain Self-Management Intervention). Remaining differences due to measure not being completed by child.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
units on a scale
  T1 (baseline): number analyzed (Participants) | 50 | 50
  T1 (baseline) | 2.7 (2.6) | 3.3 (2.7)
  T2 (12 weeks): number analyzed (Participants) | 37 | 32
  T2 (12 weeks) | 2.6 (2.5) | 3.3 (2.8)
  T3 (26 weeks): number analyzed (Participants) | 39 | 38
  T3 (26 weeks) | 2.9 (2.5) | 2.1 (2.3)

2. Primary Outcome: Pain Diary - Average Daily Activity Limitations
Description: App diary using Child Activity Limitations Inventory 9-items to measure activity limitations for 7 days Scores range from 0-100 where higher scores mean a worse outcome
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T1 (baseline): number analyzed (Participants) | 50 | 50
  T1 (baseline) | 14.1 (18.2) | 13.2 (13.1)
  T2 (12 weeks): number analyzed (Participants) | 37 | 32
  T2 (12 weeks) | 14.8 (16.6) | 10.6 (12.3)
  T3 (26 weeks): number analyzed (Participants) | 39 | 38
  T3 (26 weeks) | 12.9 (16.7) | 9.0 (12.5)

3. Primary Outcome: Adaptive Coping - Coping Attempts
Description: Coping Strategies Questionnaire for Sickle Cell Disease - Coping Attempts Factor Scores range from 0 - 180, higher scores mean a better outcome
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T1 (baseline) | 78.9 (28.8) | 79.6 (23.0)
  T2 (12 weeks): number analyzed (Participants) | 46 | 46
  T2 (12 weeks) | 83.3 (31.1) | 88.9 (27.6)
  T3 (26 weeks): number analyzed (Participants) | 46 | 47
  T3 (26 weeks) | 73.9 (28.7) | 85.7 (24.0)

4. Secondary Outcome: Treatment Acceptability
Description: Treatment Evaluation Inventory scores range from 9 - 45 where higher scores mean a better outcome
Time Frame: 2 months after starting treatment
Population: At Post-Treatment 9 subjects (4 Education Control and 5 Pain Self-Management Intervention) declined to participate or could not be reached. At Follow-up 13 subjects declined to participate or could not be reached (5 Education Control and 8 Pain Self-Management Intervention).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Child: Children in the Pain Self-Management Intervention
- Parent: Caregivers in the Pain Self-Management Intervention
Arm/Group | Child | Parent
Number analyzed (Participants) | 49 | 44
score on a scale | 34.6 (7.7) | 34.7 (5.5)

5. Secondary Outcome: Physical and Emotional Functioning - Depressive Symptoms
Description: Patient-reported Outcomes Measurement Information System (PROMIS) Pediatric Profile v2.0 - Depressive Symptoms T-score, higher scores means higher depressive symptoms. 50 indicates the population mean with a standard deviation of 10. A T-score of 60 is indicative of sub-clinical or elevated levels of depressive symptoms.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
T-score
  T1 (baseline) | 52.4 (11.5) | 49.7 (9.3)
  T2 (12 weeks): number analyzed (Participants) | 44 | 45
  T2 (12 weeks) | 52.3 (12.1) | 50.8 (9.5)
  T3 (26 weeks): number analyzed (Participants) | 46 | 46
  T3 (26 weeks) | 52.4 (11.6) | 49.3 (9.3)

6. Secondary Outcome: Physical and Emotional Functioning - Anxiety
Description: Patient-reported Outcomes Measurement Information System (PROMIS) Pediatric Profile v2.0 - Anxiety T-score, higher scores means higher levels of anxiety. 50 indicates the population mean with a standard deviation of 10. A T-score of 60 is indicative of sub-clinical or elevated levels of anxiety.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
T-score
  T1 (baseline) | 50.1 (12.2) | 50.5 (11.1)
  T2 (12 weeks): number analyzed (Participants) | 44 | 45
  T2 (12 weeks) | 50.3 (11.9) | 48.6 (10.8)
  T3 (26 weeks): number analyzed (Participants) | 46 | 46
  T3 (26 weeks) | 49.9 (11.4) | 46.9 (11.6)

7. Secondary Outcome: Physical and Emotional Functioning - Mobility
Description: Patient-reported Outcomes Measurement Information System (PROMIS) Pediatric Profile v2.0 - Mobility T-score, higher scores means better mobility. 50 indicates the population mean with a standard deviation of 10. A T-score of 40 is indicative of sub-clinical mobility limitations.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
T-score
  T1 (baseline) | 44.2 (10.3) | 42.8 (10.2)
  T2 (12 weeks): number analyzed (Participants) | 44 | 45
  T2 (12 weeks) | 43.0 (9.8) | 43.2 (9.4)
  T3 (26 weeks): number analyzed (Participants) | 46 | 46
  T3 (26 weeks) | 44.2 (9.9) | 45.4 (8.9)

8. Secondary Outcome: Physical and Emotional Functioning - Pain Interference
Description: Patient-reported Outcomes Measurement Information System (PROMIS) Pediatric Profile v2.0 - Pain Interference T-score, higher scores means more pain interference. 50 indicates the population mean with a standard deviation of 10. A T-score of 60 is indicative of sub-clinical or elevated levels of pain interference.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
T-score
  T1 (baseline) | 59.9 (12.7) | 60.0 (10.8)
  T2 (12 weeks): number analyzed (Participants) | 44 | 45
  T2 (12 weeks) | 59.2 (11.7) | 57.1 (8.9)
  T3 (26 weeks): number analyzed (Participants) | 46 | 46
  T3 (26 weeks) | 58.6 (12.7) | 54.7 (11.2)

9. Secondary Outcome: Physical and Emotional Functioning - Fatigue
Description: Patient-reported Outcomes Measurement Information System (PROMIS) Pediatric Profile v2.0 - Fatigue T-score, higher scores means higher levels of fatigue. 50 indicates the population mean with a standard deviation of 10. A T-score of 60 is indicative of sub-clinical or elevated levels of fatigue.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scaleT-score
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scaleT-score
  T1 (baseline) | 54.5 (13.7) | 57.2 (10.6)
  T2 (12 weeks): number analyzed (Participants) | 44 | 45
  T2 (12 weeks) | 55.5 (12.9) | 54.8 (11.4)
  T3 (26 weeks): number analyzed (Participants) | 46 | 46
  T3 (26 weeks) | 57.3 (11.5) | 53.2 (12.6)

10. Secondary Outcome: Physical and Emotional Functioning - Peer Relationships
Description: Patient-reported Outcomes Measurement Information System (PROMIS) Pediatric Profile v2.0 - Peer Relationships T-score, higher scores means better peer relationships. 50 indicates the population mean with a standard deviation of 10. A T-score of 40 is indicative of sub-clinical or reduced quality of peer relationships.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
T-score
  T1 (baseline) | 44.4 (10.2) | 49.2 (9.0)
  T2 (12 weeks): number analyzed (Participants) | 44 | 45
  T2 (12 weeks) | 43.3 (11.3) | 45.4 (9.1)
  T3 (26 weeks): number analyzed (Participants) | 46 | 46
  T3 (26 weeks) | 43.0 (11.0) | 46.6 (10.4)

11. Secondary Outcome: Patient Global Impression of Change
Description: Global rating for improvement in pain and functioning Scores range from 1-7 where higher scores mean a better outcome
Time Frame: 12 weeks and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T2 (12 weeks): number analyzed (Participants) | 45 | 44
  T2 (12 weeks) | 3.9 (1.8) | 4.1 (1.5)
  T3 (26 weeks): number analyzed (Participants) | 45 | 46
  T3 (26 weeks) | 3.7 (1.6) | 4.0 (1.8)

12. Secondary Outcome: Parent Protectiveness
Description: Adult Responses to Children's Symptoms Scores range from 0-4 where higher scores mean a worse outcome
Time Frame: Baseline,12 weeks, and 26 weeks
Population: At Post-Treatment 9 subjects (4 Education Control and 5 Pain Self-Management Intervention) declined to participate or could not be reached. At Follow-up 13 subjects declined to participate or could not be reached (5 Education Control and 8 Pain Self-Management Intervention). Remaining differences due to measure not being completed by parent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T1 (baseline): number analyzed (Participants) | 49 | 54
  T1 (baseline) | 2.1 (0.9) | 1.8 (0.9)
  T2 (12 weeks): number analyzed (Participants) | 41 | 42
  T2 (12 weeks) | 1.9 (0.9) | 1.5 (0.7)
  T3 (26 weeks): number analyzed (Participants) | 43 | 39
  T3 (26 weeks) | 1.7 (0.8) | 1.5 (0.9)

13. Secondary Outcome: Health Services Utilization
Description: Client Services Receipt Inventory adapted for sickle cell disease - Number of hospitalizations and/or ED visits
Time Frame: Baseline and 26 weeks
Population: At Follow-up 13 subjects declined to participate or could not be reached (5 Education Control and 8 Pain Self-Management Intervention). Remaining differences due to measure not being completed by parent.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
visits
  T1 (baseline): number analyzed (Participants) | 50 | 54
  T1 (baseline) | 2.9 (3.6) | 4.0 (4.2)
  T3 (26 weeks): number analyzed (Participants) | 43 | 39
  T3 (26 weeks) | 3.3 (4.3) | 2.5 (3.3)

14. Secondary Outcome: Parent Psychological Distress
Description: Symptom Checklist 90 - Global Severity Index Scores range from 0-4, with higher scores indicating a worse outcome
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T1 (baseline): number analyzed (Participants) | 49 | 53
  T1 (baseline) | 0.59 (0.67) | 0.41 (0.46)
  T2 (12 weeks): number analyzed (Participants) | 41 | 43
  T2 (12 weeks) | 0.51 (0.50) | 0.33 (0.39)
  T3 (26 weeks): number analyzed (Participants) | 44 | 39
  T3 (26 weeks) | 0.55 (0.52) | 0.42 (0.50)

15. Secondary Outcome: Child Physical and Emotional Functioning - Parent Report, Social Functioning
Description: Bath Adolescent Pain Questionnaire - Parent version, Social Functioning (score range: 0-36). A higher score indicates more impaired functioning for all subscales.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T1 (baseline): number analyzed (Participants) | 51 | 55
  T1 (baseline) | 12.4 (6.4) | 12.9 (6.1)
  T2 (12 weeks): number analyzed (Participants) | 44 | 43
  T2 (12 weeks) | 12.9 (5.1) | 12.4 (5.3)
  T3 (26 weeks: number analyzed (Participants) | 45 | 41
  T3 (26 weeks | 12.9 (4.8) | 13.7 (5.7)

16. Secondary Outcome: Child Physical and Emotional Functioning - Parent Report, Physical Functioning
Description: Bath Adolescent Pain Questionnaire - Parent version Physical Functioning (0-36). A higher score indicates more impaired functioning for all subscales.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T1 (baseline): number analyzed (Participants) | 49 | 55
  T1 (baseline) | 8.4 (4.2) | 10.3 (6.2)
  T2 (12 weeks): number analyzed (Participants) | 43 | 43
  T2 (12 weeks) | 10.2 (4.4) | 9.7 (4.5)
  T3 (26 weeks): number analyzed (Participants) | 44 | 41
  T3 (26 weeks) | 10.3 (5.7) | 9.7 (4.8)

17. Secondary Outcome: Child Physical and Emotional Functioning - Parent Report, Depression
Description: Bath Adolescent Pain Questionnaire - Parent version, Depression (0-24). A higher score indicates more impaired functioning for all subscales.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T1 (baseline): number analyzed (Participants) | 49 | 55
  T1 (baseline) | 7.4 (4.9) | 6.8 (4.2)
  T2 (12 weeks): number analyzed (Participants) | 43 | 43
  T2 (12 weeks) | 7.6 (4.3) | 6.5 (3.6)
  T3 (26 weeks): number analyzed (Participants) | 44 | 41
  T3 (26 weeks) | 7.3 (4.5) | 7.7 (4.2)

18. Secondary Outcome: Child Physical and Emotional Functioning - Parent Report, General Anxiety
Description: Bath Adolescent Pain Questionnaire - Parent version, General Anxiety (0-28). A higher score indicates more impaired functioning for all subscales.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T1 (baseline): number analyzed (Participants) | 49 | 55
  T1 (baseline) | 6.7 (5.0) | 7.4 (5.3)
  T2 (12 weeks): number analyzed (Participants) | 43 | 43
  T2 (12 weeks) | 7.8 (4.5) | 7.0 (4.9)
  T3 (26 weeks): number analyzed (Participants) | 44 | 41
  T3 (26 weeks) | 7.4 (5.1) | 8.8 (5.3)

19. Secondary Outcome: Child Physical and Emotional Functioning - Parent Report, Pain Specific Anxiety
Description: Bath Adolescent Pain Questionnaire - Parent version, Pain Specific Anxiety (0-28). A higher score indicates more impaired functioning for all subscales.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T1 (baseline): number analyzed (Participants) | 49 | 55
  T1 (baseline) | 12.7 (6.3) | 12.2 (6.6)
  T2 (12 weeks): number analyzed (Participants) | 42 | 43
  T2 (12 weeks) | 12.9 (6.6) | 11.1 (5.6)
  T3 (26 weeks): number analyzed (Participants) | 44 | 41
  T3 (26 weeks) | 11.5 (6.5) | 10.8 (5.4)

20. Secondary Outcome: Child Physical and Emotional Functioning - Parent Report, Family Functioning
Description: Bath Adolescent Pain Questionnaire - Parent, Family Functioning (0-48). A higher score indicates more impaired functioning for all subscales.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T1 (baseline): number analyzed (Participants) | 49 | 55
  T1 (baseline) | 13.5 (8.0) | 13.4 (7.1)
  T2 (12 weeks): number analyzed (Participants) | 42 | 43
  T2 (12 weeks) | 13.5 (6.4) | 12.9 (6.5)
  T3 (26 weeks): number analyzed (Participants) | 44 | 41
  T3 (26 weeks) | 13.2 (7.1) | 12.9 (7.7)

21. Secondary Outcome: Child Physical and Emotional Functioning - Parent Report, Development
Description: Bath Adolescent Pain Questionnaire - Parent version, Development (0-44). A higher score indicates more impaired functioning for all subscales.
Time Frame: Baseline,12 weeks, and 26 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
score on a scale
  T1 (baseline): number analyzed (Participants) | 49 | 55
  T1 (baseline) | 15.0 (8.0) | 15.7 (7.6)
  T2 (12 weeks): number analyzed (Participants) | 42 | 43
  T2 (12 weeks) | 15.3 (7.9) | 14.5 (8.6)
  T3 (26 weeks): number analyzed (Participants) | 44 | 41
  T3 (26 weeks) | 15.5 (7.5) | 14.7 (9.4)

22. Secondary Outcome: Treatment Experiences - Child
Description: Self report of treatment experiences. The number of participants with high levels of increased stress or anxiety will be reported.
Time Frame: 12 weeks and 26 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Education Control | Pain Self-Management Intervention
Number analyzed (Participants) | 54 | 57
Participants
  T2 (12 weeks): number analyzed (Participants) | 50 | 52
  T2 (12 weeks) | 1 | 0
  T3 (26 weeks): number analyzed (Participants) | 49 | 49
  T3 (26 weeks) | 2 | 0

ADVERSE EVENTS:
Time Frame: Through study completion and follow-up (average of 10 months)
Description: Stress and anxiety at a level commensurate with participation in routine activities was not considered an Adverse Event.
Arm/Group | Education Control | Pain Self-Management Intervention
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/57
Other Adverse Events (participants affected / at risk) | 0/54 | 0/57

LIMITATIONS AND CAVEATS:
Our trial recruitment and data collection spanned dates from before the COVID-19 pandemic to during the pandemic. This factor had an impact on our ability to reach our target enrollment into the trial as well as potential effects on outcome measurement.

Despite the strength of our high retention rate in the trial, we had a high level of missingness for some outcome data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03201874/Prot_SAP_000.pdf